CLINICAL TRIAL: NCT03618108
Title: Phase IIa Prospective Study to Evaluate the Safety and Measure Efficacy of Anti-chlamydophila Antibiotic Combination (ACAC) Therapy Comprising 100mg Doxycycline, 500mg Azithromycin and 300mg Rifabutin in the Treatment of Patients With Coronary Heart Disease (CHD)
Brief Title: Anti-chlamydophila Antibiotic Combination Therapy in the Treatment of Patients With Coronary Heart Disease
Acronym: ACAC-CHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19
Sponsor: Cadrock Pty. Ltd. (Other)
Collaborators: Centre for Digestive Diseases, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC10/C01
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Coronary Heart Disease; Chlamydophila Pneumoniae Infections
MeSH Terms: conditions — Coronary Disease | interventions — Doxycycline; Azithromycin; Rifabutin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical placebo capsule dosing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Subjects will be given oral capsules containing the active comparators 50mg oral capsule doxycycline, 250mg oral capsule azithromycin and 150mg oral capsule rifabutin daily (days 1 to 7). From days 8 to 90 subjects will be given 50mg oral capsule doxycycline, 250mg oral capsule azithromycin and 150mg oral capsule rifabutin twice daily.
  Interventions: Drug: Doxycycline Capsule; Drug: Azithromycin Capsule; Drug: Rifabutin Oral Capsule
- Placebo (Placebo Comparator): subjects will be given sugar capsules identical in form and size to the active comparators, 1 capsule of each bottle (3 separate capsules) daily (days 1 to 7), 1 capsule of each bottle (3 separate capsules) twice daily (days 8 to 90).
  Interventions: Drug: Placebo oral capsule; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Doxycycline Capsule — doxycycline capsule
  Other Names: Vibramycin
  Arms: Active
Drug: Azithromycin Capsule — azithromycin capsule
  Other Names: zithromax
  Arms: Active
Drug: Rifabutin Oral Capsule — rifabutin capsule
  Other Names: mycobutin
  Arms: Active
Drug: Placebo oral capsule — Placebo oral capsule identical in size and form to doxycycline
  Arms: Placebo
Drug: Placebo Oral Tablet — Placebo oral capsule identical in size and form to azithromcyin
  Arms: Placebo
Drug: Placebo oral capsule — Placebo oral capsule identical in size and form to rifabutin
  Arms: Placebo

SUMMARY:
The purpose of the study is to see whether the antibiotic combination of 100mg doxycycline, 500mg azithromycin and 300mg rifabutin is a safe and effective treatment for coronary artery disease which has not responded to 'standard treatment'.

Coronary artery disease is the process of plaque build up within the walls of the arteries responsible for supplying the heart with oxygen and nutrients. plaque is usually made up of fatty deposits, minerals and various amounts of tissue and white cells which eventually narrows the artery, reducing blood flow to the heart. The resulting damage and build up of fat leads to inflammation of the arterial wall and eventually the arteries narrow. The researchers involved in this study consider that a pathogen called Chlamydophila pneumoniae, which can live inside cells may cause this inflammation of the arterial wall.

The purpose of this study is to see if treatment with this antibiotic combination in patients with CHD is safe and effective in reducing disease severity measured at coronary angiography and improving quality of life. Approximately 60 patients will be involved in this trial. the treatment period is 90 days with a further 90 day follow up period.

DETAILED DESCRIPTION:
Chlamydophila pneumoniae has been evaluated as one potential underlying cause of CHD. The strongest evidence supporting this hypothesis comes from multiple investigators who enrolled over 19,217 subjects in 'Anti-Chlamydia trials'. However, these studies can be questioned on the basis of the type and duration of therapy. The recent change of the genus no longer permits treatment of C. pneumoniae as if it were Chlamydia trachomatis - which can generally be cured with a short course of macrolides [azithromycin, roxithromycin or clarithromycin] used in the majority of subjects analysed in this meta-analysis. C. pneumoniae is largely intra-cellular and its preferred locations (arterial muscle cells and macrophages) may contribute to its persistence in the body. C. pneumoniae can be refractory to antibiotic treatment in spite of in vitro susceptibility to various macrolides and ansamycins likely due to the use of sub-optimal dosages, which has been shown to encourage or induce persistence of C. pneumoniae in vitro. Rupp et al (2009) reported C. pneumoniae to infiltrated poptotic neutrophils that are subsequently taken up by monocyte-derived macrophages, thereby preventing clearance by the body's immune system and preventing susceptibility in the presence of antibiotics.

The previously reported trials have used short-term or recurrent treatment. The rationale for combined antibiotic long-term therapy stems from experience with other intracellular bacteria e.g. Mycobacterium tuberculosis, characterized by its dormant forms and affinity for developing resistance. The presence of infection in arterial cells with associated fibrosis and calcification for a considerable time may warrant prolonged treatment to enable antibiotic penetration into infected spaces. The occurrence of dormant forms also requires long-term treatment to anticipate the 'awakening' of dormant bacterial cells so that antibiotics can be effective during their division phase. The use of a combination therapy rather than a single agent to address dormant forms is concurrent with experience with other chronic and multiple resistant strain infections such as H. pylori, M. tuberculosis, and Mycobacterium avium paratuberculosis which are treated with combination antibiotics to minimise the development of resistant strains. Indeed, in the C. pneumoniae/CHD trials, the only trial that showed marked improvement in primary end points was the trial that used multiple antibiotics albeit for 7 days22. Hence, it would be reasonable to trial an appropriate multiple-antibiotic regimen in CHD

In this trial, antibiotics against C. pneumoniae known to be active within cells will be used. The three drugs will be administered simultaneously to minimise resistance development, and these will be used for a minimum of 3 months. At this stage ideal duration of treatment is not known.

In preliminary clinical experience of 5 subjects, with 3-6 month treatment using clarithromycin, rifabutin and doxycycline, subjects noted reduced shortness of breath, angina episodes, and marked improvement in claudication. The dosage schedule for this trial will be initiated as half doses in the first week followed by full dosages from week two onwards. This is designed as to minimize the onset of potential adverse effects in subjects. The dose-escalating schedule allows introduction of the medications into the body and maximizing bioavailability yet minimizing the potential adverse events.

The experience with long term use of a combination of three antibiotics in Mycobacterium avium paratuberculosis and Crohn's disease has been largely in younger subjects who did not receive anti-platelet agents as concomitant therapies, and thus, macrolide anti-platelet agent interactions have not been observed. In the proposed group of subjects with CHD disease, clarithromycin has a known interaction with anti-platelet agents and therefore in this group, clarithromycin will be substituted by azithromycin, a similar macrolide that demonstrates the same intracellular activity against C. pneumoniae but does not exhibit such interaction with anti-platelet agents. The azithromycin dose will be reduced due to its longer half-life, resulting in longer bioavailability duration in the body. Due to reported occasional QT-prolongation at high doses of azithromycin, ECG monitoring of the QT-interval will be carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females (without childbearing potential as evidenced by hysterectomy, tubal ligation or at least one year post-menopause) aged 18 to 80 years inclusive.
2. Ability to provide written informed consent to participate in the study.
3. Subjects with documented recent acute coronary syndrome (ACS) or evidence of myocardial ischemia.
4. Subjects who have a culprit lesion suitable for PCI, and a non-critical lesion in another vessel suitable for staged PCI with an FFR of <0.80, for subjects undergoing diagnostic angiography and FFR without ad hoc PCI.
5. No serious co-morbidities, which might interfere with the subject's ability to enter the study.
6. Able to communicate effectively with the study team and to comply with the protocol.

Exclusion Criteria:

1. Females that are of child bearing potential
2. Subjects without a non-culprit lesion considered appropriate to plan a staged PCI.
3. Clinically significant haematologic, hepatic, metabolic, renal, rheumatologic, anaphylactic reactions, neurological or psychiatric disease.
4. Clinical evidence of any other disease, which might interfere with the subject's ability to enter the trial.
5. Concomitant administration of medications that may interfere with treatment as assessed by the Investigator, including allergy to any component of the therapy.
6. Concomitant administration of any medication prohibited for use during this study (e.g. colchicine)
7. Male subjects consuming greater than 60g alcohol per day, or female subjects consuming greater than 40g alcohol per day.
8. Evidence of any recent history of, or current recreational drug abuse.
9. Serious adverse reaction or hypersensitivity to therapeutic drugs.
10. Unable and to comply with the study requirements.
11. Subjects who have been involved in an experimental drug protocol within the past four weeks.

If a subject becomes pregnant during the course of the study, they will be immediately withdrawn and treated in the way least likely to harm both subject and foetus.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
To evaluate effect of antibiotic therapy through evaluation of fractional flow reserve | day 90 post initiation of treatment (Visit 3)
  to evaluate the effect of antibiotic combination therapy on objective measures of improvement in coronary flow as determined by fractional flow reserve (FFR) in subjects undergoing percutaneous coronary intervention (PCI) with non-critical lesions in non-culprit arteries

SECONDARY OUTCOMES:
Angiographic stenoses changes | Day 90 post initiation of treatment (Visit 3)
  to evaluate angiographic stenoses changes (QCA) via diagnostic angiography during ACAC trial
Major adverse Clinical events | day 90 (visit 3) and Day 180 post initiation of treatment
  To record major adverse clinical events (MACE), including death, recurrent myocardial infarction, stroke and major bleeding via investigator adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Borody, Principal Investigator — Centre for Digestive Diseases; John French, Principal Investigator — Liverpool Hospital
Locations (1):
- Liverpool hospital, Liverpool, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Falk E, Shah PK, Fuster V. Coronary plaque disruption. Circulation. 1995 Aug 1;92(3):657-71. doi: 10.1161/01.cir.92.3.657. No abstract available. PMID 7634481
- [Background] Hermus L, Lefrandt JD, Tio RA, Breek JC, Zeebregts CJ. Carotid plaque formation and serum biomarkers. Atherosclerosis. 2010 Nov;213(1):21-9. doi: 10.1016/j.atherosclerosis.2010.05.013. Epub 2010 May 19. PMID 20627248

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT03618108/Prot_SAP_000.pdf